CLINICAL TRIAL: NCT04351646
Title: Development and Assessment of Rapid Testing for SARS-CoV-2 Outbreak (DARTS)
Brief Title: Diagnostics of COVID-19/DARTS (Development and Assessment of Rapid Testing for SARS-CoV-2 Outbreak)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 2020.0075
Record Dates: First submitted 2020-04-07; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; COVID-19; coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swabs, saliva samples, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SARS-CoV-2 negative inpatients: Hospitalised adult patients with SARS-CoV-2 negative tests.
- SARS-CoV-2 positive inpatients: Hospitalised adult patients with SARS-CoV-2 positive tests.
- SARS-CoV-2 suspected or confirmed NHS staff: Suspected or proven SARS-CoV-2 positive cases amongst health care professionals and lab staff.

SUMMARY:
This project will evaluate point-of-care / point-of-need (POC/PON) tests for the detection of the novel strain of coronavirus (2019 nCoV). We are working with Mologic Ltd, who have been funded by DFID/Wellcome Trust to develop a rapid, accurate and low cost, lateral flow assay (LFA) to detect viral circulating antigens and IgM/G against SARS-CoV-2 in less than 15 minutes.

These POC/PON tests are intended for the rapid triage of patients with fever and/or cough and to identify patients likely to be immune from previous infections. In addition to this the POC/PON tests will be designed as self-tests, offering the additional benefit of enabling wide deployment in the home and community settings. In addition, we will evaluate ELISA assays, also produced by Mologic to detect IgG and IgM (and possibly IgA) against SARS-CoV-2. Comparison of antibody and antigen dynamics over time will compare with ELISA and quantitative RT-PCR.

DETAILED DESCRIPTION:
On 12 January 2020, a novel coronavirus was identified as the cause of an outbreak of unexplained pneumonia in Wuhan City, Hubei Province, China. This coronavirus was later named SARS-CoV-2, and the disease it causes COVID-19.

SARS-CoV-2 is a non-segmented, positive sense RNA virus and part of the family of coronaviruses. Similar to the Systemic Acute Respiratory Syndrome (SARS) virus, it binds to the angiotensin-converting enzyme 2 (ACE2) receptor located on type II alveolar cells and intestinal epithelia. SARS-CoV-2 can result in a severe Acute Respiratory Distress Syndrome (ARDS) which is characterised by diffuse alveolar damage and direct viral cytopathic effect on pneumocytes. Some patients who develop COVID19 may respond with a fulminant "cytokine storm" reaction.

As of 23 March 2020, a total of 374,921 COVID-19 cases have been reported in 168 countries with a total of over 16,411 deaths (case fatality amongst confirmed cases of 4.4%) (John Hopkins's Coronavirus Resource centre). Over 293,425 cases and 13,258 deaths have been reported from countries outside mainland China. The World Health Organisation (WHO) declared on the 12th of March the SARS-CoV-2 outbreak a pandemic in the context of a Public Health Emergency of International Concern (PHEIC) [4]. Europe has rapidly become the epicentre of the pandemic and in the UK, cases are increasing daily. There have been 6,724 confirmed cases in the UK as of 23 March 2020, including 190 confirmed inpatients at St George's Hospital NHS Trust (23 March 2020 , Dr. Breathnach, personal communication).

Because of the lack of a validated serological test, the actual number, and therefore the proportion, of people that develop asymptomatic infection remains unknown. This means that an accurate case fatality estimate remains elusive. Due to the rise in the number of diagnostic samples, tests are taking longer than expected. Among the foremost priorities to facilitate public health interventions is a reliable laboratory diagnosis. Prompt case ascertainment is necessary to ensure rapid and effective contact tracing, implementation of infection prevention and control measures according to WHO recommendations, and collection of relevant epidemiological and clinical information.

Because of the lack of a validated serological test, the actual number, and therefore the proportion, of people that develop asymptomatic infections remains unknown. This means that an accurate case fatality estimate remains elusive. Due to the rise of the number of samples to diagnose, tests are taking longer than expected. Among the foremost priorities to facilitate public health interventions is a reliable laboratory diagnosis. Prompt case confirmation is necessary to ensure rapid and effective contact tracing, implementation of infection prevention and control measures according to WHO recommendations, and collection of relevant epidemiological and clinical information.

The experience in China has been that around 15% of patients with confirmed infection develop severe disease and around 5% become critically ill. In the UK, a modelling analysis by the Imperial College COVID-19 Response Team suggests that even with the implementation of self-isolation measures (household quarantine and social distancing) the surge limits for both general wards and ICU beds will be exceeded 8-fold. Furthermore, a relaxation of these mitigation measures is likely to lead to a rebound of cases until there is an effective vaccine - which is not expected for some 12-18 months. We can therefore clearly expect a significant number of inpatients with COVID-19 infection in the UK in the coming months.

The SARS-CoV-2 antigen and antibody lateral flow assay (LFA) development has been led by Mologic, a company based in Bedford. We will use prototype LFA and ELISA that are ready for preliminary evaluation, and subsequently use these tests on-site to evaluate the test at POC. LFA have been developed for SARS-CoV-2 antigen detection in throat/ nose swabs and detection of IgG and IgM in blood/serum and SARS-CoV-2 antigen detection, IgG, IgM and IgA in saliva. Saliva is an exciting sample to use as it is far easier to use than blood or throat / nose swabs for potential self-testing.

Additionally, it is currently unknown why some patients develop severe COVID-19, while others affected by the same SARS-CoV-2 infection display only mild symptoms. Co-morbidities such as hypertension, kidney disease and diabetes have been linked to poorer prognosis and clinical outcomes. However, a proportion of patients of younger age and without comorbidities also develop severe disease- and there is a need for greater understanding of the immunopathogenesis of severe COVID-19 infection is important.

The use of diagnostics developed within this study will improve the management of cases of COVID-19. The LFA are rapid, easy to use and designed to be affordable globally. The rapid diagnosis of SARS-CoV-2 with antigen detection will allow patients to be rapidly triaged in hospital, GP surgeries and other places such as immigration areas. They are sufficiently cheap to be appropriate for use in low- and middle-income countries. The use of antibody detection will allow both for diagnosis of immunological response to acute infections as well as after patients have recovered later . To utilise these tests appropriately an understanding of dynamic immunopathological changes over time is necessary.

Characterisation of immune response and susceptibility and its association with viral clearance and disease progression on in large cohorts with varied disease severity is important to assist clinical risk prediction outcomes and evaluate the potential for novel immunotherapeutic interventions. Immune response characteristics may have predictive and prognostic value, with early adaptive immune responses possibly correlated with improved clinical outcomes.

ELIGIBILITY:
==INCLUSION CRITERIA =========

Negative SARS-CoV-2:

* Aged 18 years of age or over
* Negative SARS-CoV-2 result from specimen received at SWLP laboratory in SGHFT

Positive SARS-CoV-2:

* Aged 18 years of age or over
* Positive SARS-CoV-2 result from specimen received at SWLP laboratory in SGHFT
* Requires hospitalisation in SGHFT

HCP with suspected or confirmed SARS-CoV-2:

* Aged 18 years of age
* Staff member with positive SARS-CoV-2 result from specimen received at SWLP laboratory in SGHFT or suspected diagnosis of COVID-19

==EXCLUSION CRITERIA =========

Negative SARS-CoV-2:

* Aged less than 18 years
* Outpatients
* History of known immune suppression

Positive SARS-CoV-2:

* Aged less than 18 years
* Patients unlikely to survive >28 days in view of attending medical team
* Outpatients
* Anticipated transfer to another hospital within 72 hours
* History of known immune suppression

HCP with suspected or confirmed SARS-CoV-2:

* Aged less than 18 years
* History of known immune suppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients population will include inpatients ad St George Hospital Foundation Trust (SGHFT) requiring SARS-CoV-2 test.
  Health Care Professionals population will encompass staff working at St George Hospital Foundation Trust (SGHFT) during the SARS-CoV-2 outbreak who are suspected or confirmed cases of SARS-CoV-2.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
Antibody titres to SARS-CoV-2 | Day 3 post baseline samples
  Antibody titres at day 3 post baseline samples.
Antibody titres to SARS-CoV-2 | Day 5 post baseline samples
  Antibody titres at day 5 post baseline samples.
Antibody titres to SARS-CoV-2 | Day 7 post baseline samples
  Antibody titres at day 7 post baseline samples.
Antibody titres to SARS-CoV-2 | Day 10 post baseline samples
  Antibody titres at day 10 post baseline samples.
Antibody titres to SARS-CoV-2 | Days 14 post baseline samples
  Antibody titres at day 14 post baseline samples.
Antibody titres to SARS-CoV-2 | Day 28 baseline samples
  Antibody titres at day 28 post baseline samples.
Antibody titres to SARS-CoV-2 | Day 56 post baseline samples
  Antibody titres at day 56 post baseline samples.

OTHER OUTCOMES:
Antigen dynamics | Days 3, 5, 7,10 14 and 28 and 56 post baseline samples
  Viral (SARS-CoV-2) antigen dynamics over time
HLA-KIR interactions | Days 3, 5, 7,10 14 and 28 and 56 post baseline samples
  Examine HLA-KIR interactions in relation to CD8 anti-viral responses
Plasma cytokine levels | Day 7, day 14 and optionally day 28.
  Plasma levels of cytokines (e.g. IL-1, IL-6, TNF-alpha, TGF-beta) measured by Luminex multiplex and/or ELISA assays and expressed in ug/ml
Transcriptome | Day 7, day 14 and optionally day 28.
  Total RNA will be isolated then used for cDNA synthesis and amplification. Samples will undergo 100-bp DNA sequencing, sequenced reads will be aligned to a reference genome and differentially expressed genes analysed using open source software. Pathway enrichment analysis will then be performed and the Mixture of Isoforms probabilistic framework applied to assess alternative transcription events. Differential gene expression analysis will identify key genes upregulated in COVID-19 versus control subjects, and at different timepoints in the COVID-19 disease process.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Georges Hospital Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Staines HM, Kirwan DE, Clark DJ, Adams ER, Augustin Y, Byrne RL, Cocozza M, Cubas-Atienzar AI, Cuevas LE, Cusinato M, Davies BMO, Davis M, Davis P, Duvoix A, Eckersley NM, Forton D, Fraser AJ, Garrod G, Hadcocks L, Hu Q, Johnson M, Kay GA, Klekotko K, Lewis Z, Macallan DC, Mensah-Kane J, Menzies S, Monahan I, Moore CM, Nebe-von-Caron G, Owen SI, Sainter C, Sall AA, Schouten J, Williams CT, Wilkins J, Woolston K, Fitchett JRA, Krishna S, Planche T. IgG Seroconversion and Pathophysiology in Severe Acute Respiratory Syndrome Coronavirus 2 Infection. Emerg Infect Dis. 2021 Jan;27(1):85-91. doi: 10.3201/eid2701.203074. Epub 2020 Nov 30. PMID 33256890